CLINICAL TRIAL: NCT02360839
Title: The Use of FNA and FNB in the Optimization of EUS-assisted Tissue Sampling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per Hedenström (Other)
Responsible Party: Sponsor-Investigator, Per Hedenström, Dr, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Dnr 1092-11
Record Dates: First submitted 2015-01-26; First posted 2015-02-11 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early (No Intervention): Study subjects (patients) undergoing endoscopic ultrasound (with or without FNA/TCB) for clinical reasons during 2005-2011.
- Late (Other): Study subjects (patients) undergoing endoscopic ultrasound with EUS-guided sampling of various lesions for clinical reasons during 20012-2015.
  Subjects sampled with both EUS-FNA and EUS-FNB on the same lesion. Randomization on first needle order.
  Interventions: Device: EUS-guided fine needle biopsy sampling (EUS-FNB)

INTERVENTIONS:
Device: EUS-guided fine needle biopsy sampling (EUS-FNB) — Dual sampling with EUS-FNA and EUS-FNB in a randomized order.
  Arms: Late

SUMMARY:
Endoscopic ultrasound (EUS) with fine needle aspiration (FNA) for cytology and/or fine needle biopsy (FNB) for histology may be used in the diagnostic work-up of intrathoracic and intrabdominal lesion of unknown origin. Certain lesions (such as pancreatic adenocarcinoma) are often well characterized by cytology assessment of FNA-samples while others are not (such as GIST-tumors).

This study is a part observational (early study phase) and part interventional study (late study phase) on the diagnostic accuracy of EUS-assisted tissue sampling by FNA or FNB during a 10-year period on a tertiary endoscopy centre.

DETAILED DESCRIPTION:
Variables affecting the diagnostic accuracy of EUS-FNA and EUS-FNB in different cases and tumor scenarios will be studied in detail such as the influence of medical equipment used (i.e the different types and sizes of puncture needles), the experience of the endosonographers, cytopathologists and pathologists and the use of rapid on-site evaluation of cytology samples.

Each study case is reviewed post-EUS (according to the schedule precised below) regarding further diagnostic work-up, neoadjuvant treatment, surgery result, clinical follow-up, (neo)adjuvant treatment, and survival. Non-parametrical tests will be applied as the main statistical method.

ELIGIBILITY:
Inclusion Criteria:

* Referral for a diagnostic EUS

Exclusion Criteria:

* Referral for an interventional EUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2009-07; Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The cellular quality of the EUS-FNA specimens (categorical variable). | Follow up is by time of surgery (in average 2 months after EUS-FNA)
  Specimens are measured on a standardized 5-grade categorical scale - from 1 (=poor, non-diagnostic yield) to 5 (excellent, completely diagnostic yield). There is no specific unit measured (the variable is not a continuous one). The results from cytology assessment of EUS-derived tissue are compared to the final diagnosis, that is based on the subsequent surgery report. Results from FNA and FNB are regarded equally important. That is why both are treated as Primary Outcomes.
The histological quality of the EUS-FNB specimens (categorical variable). | Follow up is by time of surgery (in average 2 months after EUS-FNB)
  Specimens are measured on a standardized 5-grade categorical scale - from 1 (=poor, non-diagnostic yield) to 5 (excellent, completely diagnostic yield). There is no specific unit measured (the variable is not a continuous one). The results from pathology assessment of EUS-derived tissue are compared to the final diagnosis, that is based on the subsequent surgery report. Results from FNA and FNB are regarded equally important. That is why both are treated as Primary Outcomes.

SECONDARY OUTCOMES:
Immunohistochemistry profiling of EUS | Follow up is by time of surgery (in average 2 months after EUS)
  The immunohistochemical (IHC) profile of tumor material from EUS-samples will be compared to the immunohistochemical profile of tissue derived from surgery of the very same case (categorical variable, Yes (1) = correct IHC-profiling by EUS or No (2) = non-correct IHC-profiling by EUS).

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Sadik, Prof, Principal Investigator — Sahlgrenska University Hospital, Gothenburg
Locations (1):
- Dr Per Hedenström, Gothenburg, Sweden

REFERENCES:
- [Derived] Hedenstrom P, Demir A, Khodakaram K, Nilsson O, Sadik R. EUS-guided reverse bevel fine-needle biopsy sampling and open tip fine-needle aspiration in solid pancreatic lesions - a prospective, comparative study. Scand J Gastroenterol. 2018 Feb;53(2):231-237. doi: 10.1080/00365521.2017.1421704. Epub 2018 Jan 4. PMID 29301477